CLINICAL TRIAL: NCT05149443
Title: Move it, Move ID! A Co-created and Theory-based mHealth Intervention to Increase Physical Activity in Adolescents With Intellectual Disability
Brief Title: Move it, Move ID! Promotion of Physical Activity in Adolescents With Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FWO/11F3621N
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Physical Activity; Health Promotion; Adolescents; Intellectual Disability
MeSH Terms: conditions — Motor Activity; Intellectual Disability | interventions — Amyloid

STUDY DESIGN:
Intervention Model Description: The effectiveness of the 'Move it, Move ID'-intervention and its two different components (i.e. buddy and gamification) will be measured through an aggregated single case design, i.e. the ABAB reversal design. Rather than taking few measurements from a sample of many individuals, many measurements are taken repeatedly from the same individual(s) in ABAB reversal designs. Participants are serving as their own controls, leading to the fact that overall sample sizes are smaller than traditional RCTs without losing adequate power.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effectiveness of the Move it, Move ID app (Experimental): All participants will receive the Move it, Move ID app.
  Interventions: Behavioral: theory-based mHealth-intervention (app)

INTERVENTIONS:
Behavioral: theory-based mHealth-intervention (app) — Measuring the effect of the buddy and gamification components separately. During the A1 phase (baseline) and the A2 phase (reversal), participants will be asked not to use the 'Move it, Move ID' intervention: the app will be blocked. After an A phase, the app will be unblocked. During the B1 and B2 intervention phase, participants use the 'Move My it, Move ID' intervention only consisting of the buddycomponent. During the intervention period, adolescents and buddies are asked to wear an accelerometer. During the first AB pair we examine whether the buddy component has an effect on PA compared to no intervention. In the A2 reversal phase possible carryover effects can be measured. It will be informative to investigate whether some parts of the intervention are automatized or internalized and will still have some effect even when participants have no access to the intervention anymore (i.e. A2 phase). The study duration is 32 days; each phase will have a duration of minimum 5 days.
  Other Names: Component 1 (buddy)
Behavioral: theory-based mHealth-intervention (app) — After the first study, other participants will be recruited. In a second study, the set-up remains the same, but the A1 and A2 phase this time consist of the buddy component (i.e. control phase) and in the B1 and B2 phase the gamification component will be added. This way, we can determine whether the gamification component has an effect on PA compared to the baseline buddy component intervention.
  The study duration is 32 days for all participants. The duration of the 4 different phases of the design will vary between participants, but each phase will have a duration of minimum 5 days.
  Other Names: Component 1+2 (buddy+gamification)

SUMMARY:
The aim of this study is to develop and implement an mHealth intervention focusing on the promotion of physical activity in adolescents with intellectual disability.

DETAILED DESCRIPTION:
Overweight and obesity are globally challenging health problems and major risk factors for a number of chronic diseases, including diabetes, cardiovascular diseases and cancer. Sufficient physical activity (PA) is an important protective factor in the development of overweight and obesity. Adolescents with intellectual disability (ID) report lower levels of PA and higher rates of overweight and obesity in comparison to adolescents without ID. There is a dire need to find ways to promote PA in adolescents with ID for their present and future health. However, while PA promotion in adolescents is a welldeveloped science, there is only a handful of studies dedicated to adolescents with ID. Consequently developing and designing PA promotion interventions specifically tailored to the needs of youth with ID is of the utmost importance. Currently, however, there is a real knowledge gap in terms of fundamental research on crucial intervention mechanisms to promote PA in adolescents with ID, as well as specific behaviour change theories adapted to this population. The aim of the current research project is to co-create and evaluate a theory-based mHealth intervention, which focuses on increasing PA for adolescents with ID.

The underlying framework within the intervention development is the Behaviour Change Wheel, together with a co-creation approach which is a bottom-up approach in which the target group (adolescents with ID in this case) is actively involved in the development of the intervention. The result of this approach is contextually appropriate intervention and intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with mild ID
* Dutch speaking
* Having a smartphone or tablet (or being able to use a test smartphone from the research group)
* Having enough motor skills to engage in PA

Exclusion Criteria:

* Adolescents with moderate, severe or profound ID

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 32 days (post-test)
  The primary outcome of the intervention is PA. To objectively measure PA, participants will be asked to wear an accelerometer (e.g., Axivity AX3).
  The purpose of buddies wearing an Axivity is to be able to explain effects afterwards regarding whether or not having a cooperating buddy during the intervention period. The Axivity will be worn on the wrist and is waterproof. As such, participants do not have to remove the Axivity during the intervention period countering the issue of non-wear.

SECONDARY OUTCOMES:
Engagement (with the app) | 32 days (post-test)
  Engagement will be measured through the use of subjective and objective measures. Experiential engagement will be assessed using the User Engagement Scale Short Form (UES-SF). Items will be assessed after the B2 intervention phase. In case of difficulties with literacy, buddies will be asked to help the participants fill in the questionnaire. However, research among people with ID shows that Likert scales are easily understood and meaningful to the respondents. In addition, individual semi-structured interviews (e.g.
  immediately post-intervention, so after B2) will be conducted to learn more about users' experiences of the intervention components. Behavioural engagement will be assessed via objective measures (usage data). A log data analysis will be conducted to track use patterns, including number of logins, their time spent online and the moment that a participant stops using the application (e.g. drop-out).

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided